CLINICAL TRIAL: NCT00761930
Title: Compare the Clinical Efficacy of Prototype Toothpastes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2007-GIN-04-RR
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Fluorides; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator): commercially available Fluoride toothpaste
  Interventions: Drug: Fluoride
- B (Active Comparator): fluoride/triclosan/copolymer toothpaste
  Interventions: Drug: Triclosan and fluoride
- C (Experimental): fluoride/herbal toothpaste
  Interventions: Drug: Herbal Ingredient and fluoride

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Other Names: Colgate Great Regular Flavor toothpaste
  Arms: A
Drug: Triclosan and fluoride — Brush twice daily
  Other Names: Colgate Total toothpaste
  Arms: B
Drug: Herbal Ingredient and fluoride — Brush twice daily
  Arms: C

SUMMARY:
Evaluate clinical efficacy of a prototype toothpaste on control of dental plaque gingival inflammation

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age
* Good general health
* Must sign informed consent form
* Minimum of 16 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients,
* relevant to any ingredient in the test products as determined by the dental/medical
* Professional monitoring the study.
* Dental Selection Criteria: Average full mouth GI score should be in the range of
* - 2.0. heavy plaque formers should be avoided. Target a full mouth PI
* (Quigley-Hein) to be in the range of 1.5-3.0
* If of child bearing potential and on birth control (diaphragm, birth control pills,
* Birth control implants, IUD (Intrauterine device), condoms)

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures
* Moderate or advanced periodontal disease
* 2 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that are currently affect salivary flow.
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this
* study.
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* History of allergy to common dentifrice ingredients
* Presence of an orthodontic appliance which interferes with plaque scoring.
* History of allergy to natural remedies, such as herbal ingredients
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
* Smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Ren, DDS, Principal Investigator
Locations (1):
- Eastman Dental Center - University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Pre-assignment Details: subjects were screened for meeting medical and oral health criteria. Then completed a 1 week washout period with fluoride toothpaste prior to receiving any study treatments.
Groups:
- A- Placebo Comparator: Commercially available Fluoride toothpaste (Colgate Great Regular Flavor toothpaste)
- B - Active Comparator: fluoride/triclosan/copolymer toothpaste (Colgate Total toothpaste)
- C - Experimental Toothpaste: fluoride/herbal toothpaste
Period: Overall Study
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste
Started | 34 | 34 | 35
Completed | 34 | 34 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste | Total
Number analyzed (Participants) | 34 | 34 | 35 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 34 | 34 | 34 | 102
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.2) | 42.68 (11.83) | 40.8 (11.7) | 41.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 23 | 74
  Male | 8 | 9 | 12 | 29
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 35 | 103

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque
Description: Quigley Hein Method: Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth. Plaque score= sum of all scores divided by the number of sites (teeth) scored.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste
Number analyzed (Participants) | 34 | 34 | 35
Units on a scale | 2.273 (0.328) | 1.806 (0.523) | 2.041 (0.403)
Statistical Analysis 1: Comparison: A- Placebo Comparator vs B - Active Comparator vs C - Experimental Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Primary Outcome: Gingivitis Score
Description: Gingivitis score (GI)= Units on a scale 0 to 3 (0 = no inflammation,
  1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding. GI scored=sum of GI scores divided by the number of sites (gingival gum line around the tooth)scored.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste
Number analyzed (Participants) | 34 | 34 | 35
Units on a scale | 0.942 (0.302) | 0.722 (0.369) | 0.705 (0.387)
Statistical Analysis 1: Comparison: A- Placebo Comparator vs B - Active Comparator vs C - Experimental Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANCOVA

3. Primary Outcome: Bleeding Index (EIBI)
Description: Eastman Interdental Bleeding Index Scores (EIBI) measures the number of interdental spaces that bleed, divided by number of interdental spaces studied to yield a score with a minimum of O and a maximum of 1 (0=no bleeding & 1= bleeding) The number of spots between teeth that bleed are divided by number of spots between teeth that are scored and may be expressed as a percent when multiplied by 100.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste
Number analyzed (Participants) | 34 | 34 | 35
Units on a scale | 0.325 (.246) | 0.164 (0.194) | 0.141 (0.183)
Statistical Analysis 1: Comparison: A- Placebo Comparator vs B - Active Comparator vs C - Experimental Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 7 weeks (1 week washout period + 6 week study test period)
Arm/Group | A- Placebo Comparator | B - Active Comparator | C - Experimental Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less